CLINICAL TRIAL: NCT05421663
Title: A Phase 1b/2, Multicenter, Open-label, Study of JNJ-90014496, an Autologous CD19/CD20 Bi-specific CAR-T Cell Therapy in Adult Participants With B-cell Non-Hodgkin Lymphoma
Brief Title: A Study of JNJ-90014496 in Participants With B-Cell Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 90014496LYM1001; 2023-506267-33-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2022-06-10; First posted 2022-06-16 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse
Keywords: CD20/CD19
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prizlo-Cel (Experimental): Participants will receive intravenous (IV) infusion of autologous prizlo-cel.
  Interventions: Biological: Prizloncabtagene autoleucel (Prizlo-Cel)

INTERVENTIONS:
Biological: Prizloncabtagene autoleucel (Prizlo-Cel) — Prizlo-Cel, an autologous dual targeting chimeric antigen receptor (CAR) - T cell therapy targeting Cluster of differentiation (CD)20 and CD19.
  Other Names: JNJ-90014496

SUMMARY:
This is a Phase 1b/2, multicenter, open-label, study of prizloncabtagene autoleucel (prizlo-cel), an autologous dual targeting chimeric antigen receptor (CAR) T-cell therapy targeting both cluster of differentiation (CD) CD20 and CD19, for the treatment of adult participants with relapsed or refractory (r/r) B-Cell non-Hodgkin lymphoma (B-NHL) or frontline high-risk diffuse large B-cell lymphoma (DLBCL).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be greater than or equal to (>=) 18 years of age, at the time of signing informed consent
* Tumor must be histologically confirmed cluster of differentiation (CD)19 and/or CD20 positive
* Must meet the indications for each subtype in Phase 1b as specified in protocol and Phase 2 participants must have following: Diagnosis of Large B-cell lymphoma (LBCL), Follicular large B-cell lymphoma (FLBCL), or transformation of indolent lymphoma; Received at least 2 prior lines of systemic therapy; Relapsed or refractory disease defined as 1 or more of the following: Stable disease or Progressive disease (PD) as best response to most recent anti-lymphoma therapy OR disease progression or recurrence after a partial response (PR) or complete response (CR) to most recent anti lymphoma therapy; cohort specific requirements as mentioned in protocol
* Measurable disease as defined by Lugano 2014 classification
* Eastern cooperative oncology group (ECOG) performance status of 0 to 2

Exclusion Criteria:

* History of symptomatic deep vein thrombosis or pulmonary embolism within six months of apheresis (line associated deep vein thrombosis is allowed)
* History of stroke, unstable angina, myocardial infarction, congestive heart failure New York Heart Association (NYHA) Class III or IV, severe cardiomyopathy or ventricular arrhythmia requiring medication or mechanical control within 6 months of apheresis
* History of a seizure disorder, dementia, cerebellar disease or neurodegenerative disorder
* Known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system
* Current active liver or biliary disease (except for Gilbert's syndrome or asymptomatic gallstones)
* Evidence of active viral or bacterial infection requiring systemic antimicrobial therapy, or uncontrolled systemic fungal infection
* Diagnosis of Human herpes virus (HHV) 8-positive DLBCL or T cell/histiocyte-rich large B-cell lymphoma or Burkitt and high-grade B-cell lymphoma with 11q aberrations (previously Burkitt-like lymphoma) or Richter's transformation or Lymphomatoid granulomatosis or Plasmablastic lymphoma or Waldenstrom's Macroglobulinemia
* Any prior solid organ or allogeneic stem cell transplantation
* Autologous stem cell transplant within 12 weeks of apheresis; Prior CAR-T cell therapy within 12 weeks of apheresis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 439 (Estimated)
Dates: Start 2022-08-12 (Actual); Primary Completion 2028-12-29 (Estimated); Study Completion 2029-03-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1b: Occurrence of Adverse Events (AEs) [Safety and Tolerability] | Up to 2 Years post prizlo-cel infusion
  Occurrence of any AEs, including dose limiting toxicities (DLTs).
Phase 2: Overall Response (OR) As Assessed by Independent Review Committee (IRC) | Up to 2 Years post prizlo-cel infusion
  Overall response is defined as a PR or CR at any point between the time of prizlo-cel infusion until PD or start of subsequent anti-lymphoma therapy, whichever occurs first (per Lugano 2014 guidelines).

SECONDARY OUTCOMES:
Phase 1b: Overall Response (OR) | Up to 2 Years post prizlo-cel infusion
  Overall response is defined as a PR or CR at any point between the time of prizlo-cel infusion until PD or start of subsequent anti-lymphoma therapy, whichever occurs first (per Lugano 2014 guidelines).
Phase 1b: Duration of Response (DOR) | Up to 2 Years post prizlo-cel infusion
  DOR is defined as the time from the first documented CR or PR after prizlo-cel infusion until PD or death, whichever occurs first (per Lugano 2014 guidelines).
Phase 1b: Pharmacokinetic Evaluation of Prizlo-Cel | Up to 2 Years post prizlo-cel infusion
  Prizlo-cel blood levels will be reported.
Phase 2: Occurrence of Adverse Events (AEs) by Severity | Up to 2 Years post prizlo-cel infusion
  Severity of AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 as follows: Grade 1 (Mild), Grade 2 (Moderate), Grade 3 (Severe), Grade 4 (Life-threatening ), Grade 5 (Death). Cytokine release syndrome (CRS), Immune effector cell-associated neurotoxicity syndrome (ICANS), and Immune effector cell-associated hemophagocytic lymphohistiocytosis-like syndrome (IEC-HS) will be graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading.
Phase 2: Complete Response (CR) | Up to 2 Years post prizlo-cel infusion
  A CR is defined as at any point between the date of prizlo-cel infusion until PD or start of subsequent anti-lymphoma therapy, whichever occurs first.
Phase 2: Duration of Response (DOR) | Up to 2 Years post prizlo-cel infusion
  DOR is defined as the time from the first documented CR or PR after prizlo-cel infusion to relapse or death, whichever occurs first.
Phase 2: Progression Free Survival (PFS) | Up to 2 Years post prizlo-cel infusion
  PFS is defined as the time from the date of prizlo-cel infusion to the date of first documented disease progression, or death due to any cause, whichever occurs first.
Phase 2: Overall Survival (OS) | Up to 2 Years post prizlo-cel infusion
  OS is defined as the time from the date of prizlo-cel infusion to the date of death due to any cause.
Phase 2: Maximum Observed Blood Concentration (Cmax) for Prizlo-Cel | Up to 2 Years post prizlo-cel infusion
  Blood samples will be analyzed to report Cmax for prizlo-cel.
Phase 2: Time to Reach Maximum Observed Cmax (Tmax) for Prizlo-Cel | Up to 2 Years post prizlo-cel infusion
  Blood samples will be analyzed to report Tmax for prizlo-cel.
Phase 2: Area Under the Blood Concentration Time Curve (AUC) for Prizlo-Cel | Up to 2 Years post prizlo-cel infusion
  AUC for prizlo-cel will be reported.
Change From Baseline of the Functional Assessment of Cancer Therapy-Lymphoma (FACT-Lym) Symptom Score | From Baseline Up to 18 months
  The FACT-Lym was developed for adult patients with lymphoma. The FACT Lym is self-administered, with a recall period for all items being the past 7 days. Responses are rated on a 5-point Likert response scale ranging from 0 "not at all" to 4 "very much". Higher scores indicate fewer symptoms and better well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (31):
- United States (13):
  - City of Hope, Duarte, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Northwestern University, Chicago, Illinois
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Rutgers Cancer Institute of New Jersey, Piscataway, New Jersey
  - Levine Cancer Institute, Charlotte, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - St. David's South Austin Medical Center, Austin, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Swedish Cancer Institute, Seattle, Washington
- Australia (4):
  - St Vincents Hospital Melbourne, Fitzroy
  - The Alfred Hospital, Melbourne
  - Fiona Stanley Hospital, Murdoch
  - Calvary Mater Newcastle Hospital, Waratah
- Princess Margaret Cancer Centre University Health Network, Toronto, Ontario, Canada
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
- Netherlands (2):
  - Erasmus MC, Rotterdam
  - UMC Utrecht, Utrecht
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (4):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - ICO L'Hospitalet - Hospital Duran i Reynals, Barcelona
  - Hosp Univ Fund Jimenez Diaz, Madrid
- United Kingdom (2):
  - University College London Hospitals, London
  - The Christie NHS Foundation Trust Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency